CLINICAL TRIAL: NCT04569383
Title: An Open, Single-center Phase I Trial to Assess the Safety, Tolerability and Immunogenicity of Two Ascending Doses of the Candidate Vaccine MVA-SARS-2-S and Heterologous Booster Vaccinations With a Licensed Vaccine Against COVID-19
Brief Title: Safety and Immunogenicity of the Candidate Vaccine MVA-SARS-2-S and a Booster Vaccination With a Licensed Vaccine Against COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: German Center for Infection Research (Other); Philipps University Marburg (Other); Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UKE-DZIF-SARS-CoV-2
Record Dates: First submitted 2020-09-21; First posted 2020-09-29 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Covid19
Keywords: MVA; vaccine; SARS-CoV-2; mRNA vaccine; heterologous
MeSH Terms: conditions — COVID-19 | interventions — BNT162 Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1x10E7 IU (low dose) (Experimental): 1x10E7 IU MVA-SARS-2-S. Subgroup will receive additionally Comirnaty
  Interventions: Biological: MVA-SARS-2-S vaccinations (days 0 & 28); Biological: Comirnaty
- 1x10E8 IU (high dose) (Experimental): 1x10E8 MVA-SARS-2-S. Subgroup will receive additionally Comirnaty
  Interventions: Biological: MVA-SARS-2-S vaccinations (days 0 & 28); Biological: Comirnaty

INTERVENTIONS:
Biological: MVA-SARS-2-S vaccinations (days 0 & 28) — Vaccination with MVA-SARS-2-S in two escalating dose regimens
Biological: Comirnaty — Vaccination with Comirnaty (21 day interval)

SUMMARY:
In this phase I first-in-human clinical trial, healthy volunteers in two different dose cohorts will be vaccinated twice with the candidate vaccine MVA-SARS-2-S. A subgroup will receive a heterologous booster vaccination with a licensed COVID-19 vaccine.

The aim of the study is to assess the safety and tolerability of the candidate vaccine and to characterize its immunogenicity.

DETAILED DESCRIPTION:
The vaccine contains a Modified Vaccinia Virus Ankara (MVA) vector expressing the SARS-CoV-2 spike protein (S). A total of 30 participants will receive the following vaccine regime:

15 participants will receive 10^7 infectious units (IU) of MVA-SARS-2-S on days 0 and 28.

15 participants will receive 10^8 IU of MVA-SARS-2-S on days 0 and 28. Safety and immunogenicity data will be collected throughout the study, which concludes at day 168.

A subgroup will receive a heterologous booster vaccination with a licensed COVID-19 vaccine. Vaccinees will receive two doses of the Comirnaty vaccine (21 days interval).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Healthy male and female adults aged 18-55 years
* No clinically significant health problems as determined during medical history and physical examination at screening visit
* Body mass index 18.5 - 30.0 kg/m2 and weight > 50 kg at screening
* Adults male or non-pregnant, non-lactating female with negative pregnancy test
* Males and females who agree to comply with the applicable contraceptive requirements of the protocol

Inclusion criteria for the subjects before the 3rd/4th (=booster) vaccination:

1. Ability to understand the subject information and to personally name, sign and date the in-formed consent to participate in the study.
2. Provided written informed consent.
3. Continues to be in stable health condition as determined during medical history and physi-cal examination on vaccination visits.
4. Non-pregnant, non-lactating female with a negative pregnancy test at screening and on dosing days (prior to vaccination).
5. Be willing to refrain from blood donation during the course of the study.
6. The subject is co-operative and available for the entire study.
7. Need to have participated in previous part of the MVA-SARS-2-S vaccine study (Eudra-CT No: 2020-002998-10)

Exclusion Criteria:

* Prior exposure to SARS-CoV-2
* Receipt of any vaccine from 4 weeks prior to each trial vaccination (8 weeks for live vaccines) to 6 weeks after each trial vaccination
* Previous rMVA immunization
* Known allergy to the components of the SARS-CoV-2 vaccine product
* Known history of anaphylaxis to vaccination or any allergy likely to be exacerbated by any component of the trial vaccine
* Evidence in the subject's medical history or in the medical examination that might influence either the safety of the subject or the absorption, distribution, metabolism or excretion of the investigational product
* Clinically relevant findings in ECG
* Any confirmed or suspected immunosuppressive or immunodeficient condition, cytotoxic therapy in the previous 5 years, and/or diabetes
* Any chronic or active neurologic disorder, including seizures, and epilepsy, excluding a single febrile seizure as a child

Exclusion criteria for the subjects before the 3rd/4th (=booster) vaccination:

1. Prior infection with SARS-CoV-2 in medical history (documented by PCR test)
2. Receipt of any vaccine from 2 weeks prior to each trial vaccination (4 weeks for live vac-cines) to 2 weeks after each trial vaccination.
3. Receipt any COVID-19 vaccine (investigational or licensed other than MVA-SARS-2-S be-fore vaccination throughout end of study).
4. Known allergy to the components of t Comirnaty®.
5. Known history of anaphylaxis to vaccination or any allergy likely to be exacerbated by any component of the trial vaccine.
6. Participation in a clinical trial other than the MVA-SARS-2-S vaccine trial or use of an in-vestigational product other than MVA-SARS-2-S within 30 days or five times the half-life of the investigational product -whichever is longer- prior to receiving the first dose within this study.
7. Evidence in the subject's medical history or in the medical examination that might influence

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2021-08-24 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Experiencing Solicited Local or Systemic Reactogenicity as Defined by the Study Protocol | during the entire study (up to 6 months)
  Safety and reactogenicity will be assessed by observation, questionaire and diary. Occurence of Serious Adverse Events (SAE) will be collected throughout the entire study duration.

SECONDARY OUTCOMES:
Immunogenicity. Number of participants who seroconverted | during the entire study (up to 6 months)
  Magnitude of SARS-CoV2-specific antibody responses (ELISA and neutralization assays) monitored in an approved laboratory

CONTACTS AND LOCATIONS:
Overall Officials: Marylyn M Addo, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- CTC North GmbH & Co KG at the University Medical Center Hamburg-Eppendorf, Hamburg, Germany

REFERENCES:
- [Derived] Grewe I, Friedrich M, Dieck ML, Spohn M, Ly ML, Krahling V, Mayer L, Mellinghoff SC, Rottstegge M, Kraemer R, Volz A, Becker S, Fathi A, Dahlke C, Weskamm LM, Addo MM. MVA-based SARS-CoV-2 vaccine candidates encoding different spike protein conformations induce distinct early transcriptional responses which may impact subsequent adaptive immunity. Front Immunol. 2024 Dec 19;15:1500615. doi: 10.3389/fimmu.2024.1500615. eCollection 2024. PMID 39749328